CLINICAL TRIAL: NCT00259077
Title: A Double-blind, Randomised, Parallel-group, Multicentre, Phase III Study to Compare the Efficacy of Omeprazole 20mg and 10mg od for the Four-week Treatment of Non-erosive Reflux Disease (NERD) With That of Placebo od and to Investigate Safety
Brief Title: Four-week Omeprazole Treatment of Non-erosive Reflux Disease in a Japanese Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9587C00001; D9584L00002
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Non-erosive Reflux Disease
MeSH Terms: conditions — Non-Erosive Reflux Disease | interventions — Omeprazole

INTERVENTIONS:
Drug: Omeprazole

SUMMARY:
The purpose of this study is to study safety and efficacy of omeprazole standard treatment in a Japanese non-erosive reflux disease population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who identified their predominant symptom as heartburn and were classifiend as Grande M or N according to Hoshihara's modofied version of Los Angeles Classification at esophagogastroduodenoscopy.

Exclusion Criteria:

* Patients with any ongoing gastrointestinal bleeding at the time of esopgahogastroduodenoscopy, patients with any history of erosive esophagitis or any other major diseases or concommittant drugs likely to interfere with the evaluation of this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2003-10; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of omeoprazole 20mg and omeprazole 10mg by assessment of complete resolution rate of heartburn during the fourth week of treatment.

SECONDARY OUTCOMES:
Complete resolution of heartburn during the first and second week of treatment, assessment of sufficient relief rates of heartburn, assessment of nocturnal heartburn, assessment of other GERD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Medical Science Director, MD, Study Director — AstraZeneca
Locations (26):
- Japan (26):
  - Asa
  - Beppu
  - Chiyoda City
  - Fujieda
  - Fukuoka
  - Kanagawa
  - Kawagucki
  - Kita-ku
  - Kitakyushu
  - Kyoda
  - Meguro City
  - Minato
  - Mitsukaidō
  - Miyaodai
  - Nagoya
  - Nanao
  - Onoda
  - Osaka
  - Ōta-ku
  - Ōtsu
  - Sapporo
  - Shinagawa City
  - Shinjuku
  - Tokyo
  - Ube
  - Yukuhashi